CLINICAL TRIAL: NCT04852718
Title: Evaluate a Rehabilitation Program for the Sequelae of COVID 19 Infection: Description of a Clinical Practice
Brief Title: Rehabilitation Program for the Sequelae of COVID 19 Infection
Acronym: ISIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-COV-2020-155
Record Dates: First submitted 2021-04-15; First posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
SUBPROJECT 1:

Describe the situation of post-Covid patients in terms of muscle (skeletal and respiratory), cognitive, emotional and health-related quality of life in the 1st visit of the multidisciplinary post-covid rehabilitation consultation at the Hospital.

Retrospective observational study. The data collected in clinical records during the first visit in the post-covid Rehabilitation consultation will be analysed.

SUBPROJECT 2:

Evaluate the response to a personalized rehabilitation program in patients with post-covid sequelae in terms of muscle (skeletal and respiratory), and health-related quality of life.

Prospective observational study of a single cohort of patients. The data will be collected from successive clinical visits.

ELIGIBILITY:
Inclusion Criteria:

* • Patients who were diagnosed with Covid-19 pneumonia, confirmed by serological tests or molecular biology test (PCR), and who were at home at the time of the 1st visit.

  * PCR or serological negative test or more than 28 days after diagnosis.
  * Dyspnoea in activities of daily living (mMRC ≥ 2), (Annex 5 of the clinical protocol).
  * Patients who had muscle weakness (Clinical Frailty Scale ≥ 3), (Annex 1 of the clinical protocol).

Exclusion Criteria:

* Patients with disease activity.
* Live outside the reference area of the Hospital de la Santa Creu i Sant Pau.
* Patients with cognitive impairment that makes it difficult to carry out the rehabilitation program.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: • Patients who were diagnosed with Covid-19 pneumonia, confirmed by serological tests or molecular biology test (PCR), and who were at home at the time of the 1st visit.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-04-13 (Estimated); Primary Completion 2021-04-13 (Estimated); Study Completion 2021-04-13 (Estimated)

PRIMARY OUTCOMES:
Muscular function | 1 year
  Short Physical Performance Battery (SPPB) value 0-12

SECONDARY OUTCOMES:
Health-related Quality of life | 1 year
  SF36 questionnaire, vaule 0-100
Respiratory muscle function | 1 year
  Maximal inspiratory pressure (MIP) Maximal expiratory pressure (MEP)
Exercise capacity | 1 year
  Six-minute walking Test (6MWT): meters,

CONTACTS AND LOCATIONS:
Overall Officials: Maria-Rosa Güel-Rous, PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

REFERENCES:
- [Derived] Perrot JC, Segura M, Beranuy M, Gich I, Nadal MJ, Pintor A, Terra J, Ramirez E, Paz LD, Bascunana H, Plaza V, Guell-Rous MR. Comparison of post-COVID symptoms in patients with different severity profiles of the acute disease visited at a rehabilitation unit. PLoS One. 2022 Sep 16;17(9):e0274520. doi: 10.1371/journal.pone.0274520. eCollection 2022. PMID 36112577